CLINICAL TRIAL: NCT02148289
Title: Dietary Nitrate in COPD: A Double-blind, Randomized, Placebo-controlled, Crossover Trial
Brief Title: Dietary Nitrate in COPD
Acronym: CHB-BRJ-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHB-BRJ-COPD
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, beetroot, dietary nitrate, nitric oxide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beverage (Active Comparator): Nitrate rich beverage will contain 140ml nitrate rich beetroot juice + 200ml blackcurrant juice containing 12.7mmol nitrate
  Interventions: Dietary Supplement: Nitrate rich beverage
- Nitrate free beverage (Placebo Comparator): Nitrate free beverage will 140ml water + 200ml blackcurrant juice containing <0.5mmol nitrate
  Interventions: Dietary Supplement: Nitrate free beverage

INTERVENTIONS:
Dietary Supplement: Nitrate rich beverage — Following randomisation on day 1, subjects will consume either the nitrate or nitrate-free beverage and then the crossover beverage on day 8.
  Other Names: Nitrate rich beetroot juice
  Arms: Nitrate rich beverage
Dietary Supplement: Nitrate free beverage — Following randomisation on day 1, subjects will consume either the nitrate or nitrate-free beverage and then the crossover beverage on day 8.
  Other Names: Placebo beverage
  Arms: Nitrate free beverage

SUMMARY:
The acute consumption of dietary nitrate has been shown to improve exercise capacity in athletes, healthy adults and subjects with peripheral vascular disease. Many COPD patients have reduced exercise capacity, The investigators hypothesized that acute nitrate consumption, in the form of beetroot juice, might increase incremental shuttle walk test (ISWT) distance in COPD subjects.

DETAILED DESCRIPTION:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to improve exercise capacity in athletes, healthy adults and subjects with peripheral vascular disease. Many COPD patients have reduced exercise capacity, The investigators hypothesized that acute nitrate consumption might increase incremental shuttle walk test (ISWT) distance in COPD subjects compared to a matched, low-nitrate drink.

This study is a randomized, double-blind placebo-controlled, crossover trial.

Resting blood pressure, phlebotomy and ISWT are performed. Following completion, each subject is randomized to consume beetroot juice or placebo. 3 hours later, the same assessments are repeated by the same people. After a 7d washout, the entire protocol is repeated with the crossover beverage.

ELIGIBILITY:
Inclusion Criteria:

* Information consenting out-patients with a previous physician diagnosis of COPD
* Clinically stable
* Ambulatory

Exclusion Criteria:

* Subjects who required supplemental oxygen for exercise
* Subjects with pulmonary hypertension and angina
* Intolerant to beetroot
* Insulin dependent diabetes
* Thyroid disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Incremental Shuttle Walk Test Distance | day 1, time 0, day 1, time 3h, day 8, time 0, day 8, time 3h
  The change between day 1, time 0 and day 1, time 3h will be compared to the changes between day 8, time 0 and day 8, time 3h.

OTHER OUTCOMES:
Resting blood pressure | day 1, time 0, day 1, time 3h, day 8, time 0, day 8, time 3h
  The change between day 1, time 0 and day 1, time 3h will be compared to the changes between day 8, time 0 and day 8, time 3h.

CONTACTS AND LOCATIONS:
Overall Officials: Conor P Kerley, BSc, Study Director — University College Dublin; Liam J Cormican, MD, Principal Investigator — Royal College of Surgeons in Ireland